CLINICAL TRIAL: NCT06801106
Title: ACAPELLA VERSUS LUNG FLUTE in TREATMENT of CHRONIC OBSTRUCTIVE PULMONARY DISEASE
Brief Title: Acapella Versus Lung Flute in Treatment of COPD Patients the Study Aims to Identify the Preference Between the Two Devices According to Treatment of COPD Patients Regarding Pulmonary Function Tests , Exercise Tolerence and Quality of Life Questionnaire,
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health and Population, Egypt (Other Government)
Responsible Party: Principal Investigator, Ahmed Hussein El Dessouky, B.Sc. in Physical Therapy (2009) Physical Therapist at Abu El Nomros Central Hospital, Ministry of Health and Population, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002208
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2021-01

CONDITIONS: Chronic Obstructive Airway Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Acapella (Experimental): patients received medical treatment only and conventional chest physical therapy (including diaphragmatic breathing, postural drainage, vibration and huffing and coughing techniques) in addition to respiratory training using acapella device for one time day after day for 8 consecutive weeks.
  Interventions: Device: Acapella
- Lung flute (Active Comparator): patients received medical treatment only and conventional chest (including diaphragmatic breathing, postural drainage, vibration and huffing and coughing techniques) physical therapy in addition to respiratory training using Lung flute device one time day after day for 8 consecutive weeks.
  Interventions: Device: Lung flute

INTERVENTIONS:
Device: Acapella — is an airway clearance device that combines the resistive features of a positive expiratory pressure device with oscillations, which diminishes the mucus adhesiveness and decrease the collapsibility of airways
  Arms: Acapella
Device: Lung flute — is a new oscillatory positive expiratory pressure (OPEP) device that produces a low frequency acoustic wave with vigorous exhalation that increases mucociliary clearance
  Arms: Lung flute

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a prevalent and progressive condition characterized by persistent airflow limitation and chronic respiratory symptoms. Among the many approaches to managing COPD, airway clearance techniques (ACTs) play a pivotal role in improving pulmonary function, reducing symptoms, and enhancing quality of life. So, this study aimed to investigate the comparative efficacy of two ACT devices-the Acapella® and the Lung Flute®- on improving pulmonary function, exercise capacity, and quality of life in COPD patients.

The Acapella® and the Lung Flute®. Both devices utilize distinct mechanisms to facilitate mucus clearance and improve lung function. The Acapella® combines positive expiratory pressure (PEP) with oscillatory vibration, aiding in the loosening and mobilization of mucus . On the other hand, the Lung Flute® generates low-frequency sound waves through patient exhalation, stimulating mucus movement from the peripheral to central airways . While both devices have demonstrated efficacy in previous studies, there is limited comparative research evaluating their impact in COPD patients.

DETAILED DESCRIPTION:
A controlled randomized study having 70 individuals with COPD was conducted. Before the treatment began, all participants signed a permission after being informed about the study's specifics and their rights as patients. The Ethics Committee Board of Cairo University's Faculty of Physical Therapy authorized this study (P.T.REC/012/002208). The research was done in accordance with the Helsinki 0 male COPD patients aged 40-60 years, recruited from Kasr Al Ainy Hospital, Cairo University. Participants were diagnosed with moderate to severe COPD and were randomly assigned into two groups: Group A received Acapella® therapy alongside standard chest physiotherapy, and Group B received Lung Flute® therapy with the same physiotherapy protocol. Both groups underwent interventions every other day for eight weeks. Outcomes were assessed using pulmonary function tests (PFTs), the six-minute walk test (6MWT), and the VQ11 quality-of-life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

- Moderate and mild severe COPD patients were selected according GOLD guidelines.

* All patients were diagnosed as COPD with chronic bronchitis for at least two years.
* All Patients were using their prescribed medications including Broncho-dilators and mucolytics.
* Patients ceased smoking 2 months before undergoing the study.
* Patients were selected of BMI between 25-34.9.

Exclusion Criteria:

* • History of osteoporosis, significant gastro-esophageal reflux, hiatus hernia.

  * Recent acute cardiac event (6 weeks) or congestive cardiac failure.
  * Any significant musculoskeletal disorders.
  * Presence of active hemoptysis.
  * Presence of malignant disease.
  * Patients undergoing exacerbations.
  * Patients of hospital admission in last 6 month.
  * Patients with cough, rhonchi, and expectoration in last 6 month.
  * Patients who undergo exertional desaturation of oxygen below 90% after 6MWT.
  * Patients who suffer from prolonged recovery time of HR for more than one minute after finishing 6MWT.
  * Prolonged recovery time of heart rate <1 min.
  * Patients who cannot walk.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — males only
Enrollment: 70 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
• Spirometer | pulmonary functions will be measured at baseline, and it will be measured again after eight weeks.
  Spirometer will be used to assess pulmonary functions ( FEV1 , FEV 6 , FVC , FEV1/ FVC)
6 minute walk test | 6 min walk test will be measured at baseline, and it will be measured again after eight weeks
  The 6MWT measures exercise tolerance in people with various health conditions. Not only is the test a way to measure the general health of an individual, but a doctor can also use it to monitor the effectiveness of the current treatment plan and see whether it is improving a person's condition
The VQ11 Quality of life questionnaire | Vq 11 will be measured at baseline, and it will be measured again after eight weeks
  was used to determine the functional, psychological, relational and total scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt, Egypt